CLINICAL TRIAL: NCT04429139
Title: Photodynamic Therapy With Visudyne for Human Retinoblastoma: A Preliminary Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Chen-jin, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011MEKY0015
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Retinoblastoma
Keywords: Photodynamic therapy; Retinoblastoma; Visudyne; Verteporfin
MeSH Terms: conditions — Retinoblastoma | interventions — Photochemotherapy; Neoadjuvant Therapy; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PDT treatment group (Experimental): All the patients received once PDT with Visudyne® as the initial treatment. Rescue treatment with systemic chemotherapy would be given to patients if tumors were insensitive to PDT treatment, the tumors became larger, or disease relapse.
  Interventions: Drug: photodynamic therapy

INTERVENTIONS:
Drug: photodynamic therapy — PDT with Visudyne® was performed under general anesthesia according to the standard TAP study with some modifications: Verteporfin (6 mg/m2, Visudyne®; Novartis International AG, Basel, Switzerland) was injected intravenously with a standard 10-min infusion followed by followed by application of diode laser (Opal Photoactivator; Coherent Medical Group, Santa Clara, USA) (689 nm, 50 J/cm2, 600 mW/cm2) for 200 seconds to generate 120 J/cm2.
  Other Names: systemic chemotherapy; Laser photocoagulation; Cryotherapy

SUMMARY:
To study the effectiveness and safety profiles of photodynamic therapy (PDT) for the treatment of human retinoblastoma.

DETAILED DESCRIPTION:
Retinoblastoma is the commonest primary intraocular malignancy in infancy and early childhood. Ophthalmologist are trying to seek other more safe and effective treatment modalities to well control the tumor and preserve the visual function. Photodynamic therapy (PDT) is a potentially therapeutic approach for retinoblastoma which has been underestimated. In this study, we are gonging to investigate the the effectiveness and safety profiles of photodynamic therapy (PDT) for the treatment of human retinoblastoma.

ELIGIBILITY:
Inclusion Criteria:

* patients with intraocular retinoblastoma of Group A-D

Exclusion Criteria:

* (1) patients with intraocular retinoblastoma of group E; (2) patients with extraocular spread; (3); media opacities such as corneal opacity, significant cataract, or vitreous hemorrhage obscuring fundus examination; (4) patients who were allergic to verteporfin or other benzoporphyrin derivatives.

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
eye enucleation | 3 years
  the rate of eye enucleation of patients with retinoblastoma in different groups

CONTACTS AND LOCATIONS:
Locations (1):
- Kunbei Lai, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No